CLINICAL TRIAL: NCT05861622
Title: Examining the Efficacy of a Novel Moisturizer Across Eight Weeks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thu Brulé (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20257
Record Dates: First submitted 2023-04-03; First posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Skin Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Novel moisturizer (Experimental): Subjects will apply the test product twice daily, both in the morning and the evening.
  Interventions: Other: Moisturizer

INTERVENTIONS:
Other: Moisturizer — The test product is a novel moisturizer, that contains active ingredients, including rambutan extract, niacinamide, and glycoin.

SUMMARY:
Skin moisture is critical to avoid long-term skin damage. Without the necessary moisture, skin is unlikely to have the properties most commonly associated with healthy skin. Recent research has recently highlighted that rambutan extract, niacinamide, and glycoin can all help promote skin moisture and health. To help people experience better skin health, Thu Brulé has developed a serum designed to be used twice daily. Specifically, the test product in this trial was designed to help moisturize the skin and help lock in that moisture. The purpose of this trial is to examine the efficacy of the test product across an eight-week hybrid trial. The outcomes of interest include participants' perceptions of skin health and photographs/images taken of the skin.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 30-80.
* Frequently experience dry skin.
* Must experience early-stage wrinkles that are not treated by topical or oral prescription drugs/medication or over-the-counter products (e.g., Adapalene/Differin)
* Must be in good health with no unstable, uncontrolled health conditions.
* Must follow a stable, consistent dietary regimen.
* May experience hyperpigmentation and dark spots.
* Must be willing to maintain the following daily skincare routine: Daily cleansing, test product, and sunscreen that is at least SPF 30
* Must discontinue retinoids four weeks before the study start date and not use retinoids during the trial.
* Must be willing to communicate in English.
* Must be willing to use the test product as directed (twice daily)
* Must be willing to come to the Citruslabs office in Santa Monica, California at the beginning and end of the study.

Exclusion Criteria:

* Females who are pregnant or breastfeeding
* Currently participating in another research study.
* Currently using oral retinoids.
* Individuals with self-reported very oily skin.
* Individuals with cystic acne or otherwise very acne-prone skin.
* Anyone using oral acne treatments (e.g., accutane).
* Anyone prone to experiencing strong bouts of hormonal acne.
* Anyone using prescription medication relevant to the skin.
* Undergoing any cosmetic procedures during the study, including Botox, laser, or chemical peel treatments.
* Use of prescription drug (topical or oral) that is targeted at any sort of skin condition (e.g., retinoids)
* Anyone with learning and/or cognitive difficulties that prevent him/her from reading and understanding questionnaires and surveys (e.g., dementia)
* Severe chronic conditions, including oncological conditions or psychiatric disorders.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-10-13 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Perceived changes in skin health | Week 8
  Survey based assessment of participants perceived skin health. Data was collected using a textual 5-point Likert scale for each question, such as "Not noticeable" to "severe." Symptom-related questions were conducted at baseline and each check-in. The textual Likert data was transformed into numerical values of 1-6, with 6 representing the most beneficial response (i.e, "not noticeable" response to the question, "how would you rate the severity of your wrinkles") and 1 representing the least favorable/worse outcome ("severe").
Changes in skin health via VISIA® imaging | Baseline to Week 8
  VISIA® Skin Analysis system will be used to assess changes in skin outcomes. Analysis will be conducted by a board-certified dermatologist at Baseline and Week 8. The VISIA® Skin Analysis system will be used to capture the images which will then be processed by the VISIA software. The software utilizes advanced algorithms to detect and measure specific skin attributes. The skin attributes/parameters evaluated will be Wrinkles, Spots, Pores, Texture, Redness and UV Damage. These parameters are evaluated using the captured images and the specialized algorithms employed by the VISIA software. The results are then used to generate a comprehensive analysis report, which includes both the quantitative measurements and qualitative assessments, along with any corresponding scores or ratings assigned to different skin attributes. Mean participant's scores for each parameter will be calculated at Baseline and Week 8 and compared for statistical significance.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States